CLINICAL TRIAL: NCT01650688
Title: Difference in Grades of Epiblepharon According to Positional Changes and General Anesthesia
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0315
Record Dates: First submitted 2012-07-15; First posted 2012-07-26 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Epiblepharon
Keywords: Epiblepharon, general anesthesia, positional change

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epiblepharon: subjects demonstrating prominent corneal touch by cilia and/or related subjective symptoms

SUMMARY:
Epiblepharon is a very common condition among Asian children and is a fold of the skin and underlying pretarsal orbicularis muscle that overlaps the eyelid margin and pushes the lashes against the cornea. It is manifested by the anterior lamella overriding the posterior lamella which causes the lashes to brush against the cornea. Although the prevalence of epiblepharon is known to be high among Asians, its cause remains controversial. Several etiological factors may be involved in the pathogenesis of epiblepharon.

Although epiblepharon in the lower lids lessens and disappears with age in many cases, surgery must be performed at an early age in severe cases in order to prevent ocular trauma as the vertically oriented cilia of the lashes can erode the corneal epithelium. Induced keratitis and astigmatism are indications for surgical intervention.

Over our many years of surgical experience, the investigators came to realize that the severity of epiblepharon was reduced when patients were under general anesthesia during surgery. The purpose of this study was to investigate the role of the orbicularis muscle in the pathogenesis of lower lid epiblepharon and to analyze the differences in the severity of epiblepharon in the upright versus the supine position and before and after the induction of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* subjects younger than 12 years
* more than 12 months' follow-up
* subjects demonstrating prominent corneal touch by cilia and/or related subjective symptoms
* subjects who underwent general anesthesia for surgical correction of epiblepharon

Exclusion Criteria:

* subjects older than 12 years
* less than 12 months' follow-up -. subjects who underwent surgery on local anesthesia

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects with epiblepharon which needed surgical correction
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Degree of skin fold height | 1 hour before epiblepharon surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Rhiu S, Yoon JS, Zhao SY, Lee SY. Variations in the degree of epiblepharon with changes in position and induction of general anesthesia. Graefes Arch Clin Exp Ophthalmol. 2013 Mar;251(3):929-33. doi: 10.1007/s00417-012-2186-2. Epub 2012 Nov 1. PMID 23111494